CLINICAL TRIAL: NCT04163341
Title: Tailored Response to Psychiatric Comorbidity to Improve HIV Care Engagement in the United States
Acronym: TRACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael J Mugavero, MD (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor-Investigator, Michael J Mugavero, MD, Professor, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300004217
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS; Depression; Anxiety; Post-traumatic Stress Disorder; Substance Use Disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Common Elements Treatment Approach (CETA) protocol (Experimental): Adapted Common Elements Treatment Approach (CETA): The intervention is a transdiagnostic cognitive behavioral therapy approach to treating any combination of depression, anxiety, post-traumatic stress, or substance use disorder that has been adapted the needs of adults with HIV and to additionally address HIV care engagement.
  Interventions: Behavioral: Adapted Common Elements Treatment Approach
- Enhanced Usual Care (EUC) (No Intervention): Enhanced Usual Care (EUC): Usual care at the 1917 Clinic for patients with mental health concerns includes referral to a clinic social worker or counselor or to an external mental health clinic as needed. Usual care was enhanced by providing the participant's medical provider with information about the participant's elevated mental health symptoms at enrollment and recommendations for treatment.

INTERVENTIONS:
Behavioral: Adapted Common Elements Treatment Approach — The intervention is a transdiagnostic cognitive behavioral therapy approach to treating any combination of depression, anxiety, post-traumatic stress, or substance use disorder that has been adapted the needs of adults with HIV and to additionally address HIV care engagement.
  Arms: Common Elements Treatment Approach (CETA) protocol

SUMMARY:
This pilot randomized clinical trial will randomize 60 participants 1:1 to either enhanced usual care or to adapted Common Elements Treatment Approach (CETA), a counseling intervention for HIV care engagement plus depression, anxiety, PTSD, and/or substance use.

DETAILED DESCRIPTION:
Patient participants in this study will be randomized 1:1 to either enhanced usual care or the adapted CETA intervention. Enhanced usual care will include provision of feedback about psychiatric diagnoses to the HIV provider and the clinic's behavioral health team for follow-up according to the clinic's standard care. Participants randomized to the adapted CETA arm will initiate CETA with the trained counselor. The number of CETA sessions will depend on the patient's presentation but will range from 7-13 weekly in-person 1-hour sessions.Before randomization, enrolled participants will complete a baseline assessment including sociodemographic information; self-reported health; standardized assessments of depressive, anxiety, and post-traumatic stress symptoms and substance use; and key related structural and psychosocial factors including housing stability,intimate partner violence (IPV), other violence in the home, coping, social support, and experiences of stigma related to mental health.

Participants in the Enhanced Contact arm will complete a follow-up research assessment at 3 months post baseline.Participants in the adapted CETA arm will complete this assessment after the final CETA session,also expected to be at approximately 3 months post-baseline. All participants will complete a final research assessment at 9 months post-baseline (approximately 6 months post-treatment exit for those in the adapted CETA arm). These follow-up assessments will assess the same domains as the baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Patient receiving HIV care at University of Alabama at Birmingham (UAB) 1917 Clinic.
3. Elevated symptoms of depression, anxiety, post-traumatic stress, or substance use disorder: At least one of the following:

   1. Patient Health Questionnaire-9 score >= 10;
   2. Generalized Anxiety Disorder 7-Item Scale score >= 10;
   3. Post-Traumatic Stress Symptoms Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) score >= 33;
   4. ASSIST score >=11 for alcohol or >=4 for any other substance
4. At risk for suboptimal HIV care engagement: At least one of the following:

   1. Engaged in HIV care for the first time within the past 6 months;
   2. Have an HIV RNA viral load >1,000 copies/mL within the past 6 months;
   3. Antiretroviral regimen was changed due to treatment failure within the past 6 months;
   4. No-showed to an HIV primary care appointment within the past year.
5. Willing to provide written informed consent.

Exclusion Criteria:

* 1. Non-English speaking 2. Unable to attend counseling sessions 3. Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pence, PhD, Principal Investigator — UNC-Chapel Hill; Bradley Gaynes, MD, Principal Investigator — UNC-Chapel Hill; Doyane Darnell, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pence BW, Darnell D, Ranna-Stewart M, Psaros C, Gaynes BN, Grimes L, Henderson S, Parman M, Filipowicz TR, Gaddis K, Dorsey S, Mugavero MJ. Provocative Findings From a Transdiagnostic Counseling Intervention to Improve Psychiatric Comorbidity and HIV Care Engagement Among People With HIV: A Pilot Randomized Clinical Trial. J Acquir Immune Defic Syndr. 2024 Sep 1;97(1):68-77. doi: 10.1097/QAI.0000000000003457. PMID 39116333

RESULTS

PARTICIPANT FLOW:
Groups:
- CETA Protocol: Adapted Common Elements Treatment Approach: The intervention is a transdiagnostic cognitive behavioral therapy approach to treating any combination of depression, anxiety, post-traumatic stress, or substance use disorder that has been adapted the needs of adults with HIV and to additionally address HIV care engagement.
- Enhanced Usual Care: Enhanced Usual Care (EUC): Usual care at the 1917 Clinic for patients with mental health concerns includes referral to a clinic social worker or counselor or to an external mental health clinic as needed. Usual care was enhanced by providing the participant's medical provider with information about the participant's elevated mental health symptoms at enrollment and recommendations for treatment.
Period: Overall Study
Arm/Group | CETA Protocol | Enhanced Usual Care
Started | 30 | 30
Completed | 25 | 26
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CETA Protocol | Enhanced Usual Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (9.4) | 44.0 (13.4) | 41.9 (11.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 18 | 15 | 33
  Female | 10 | 12 | 22
  Transgender Male | 1 | 0 | 1
  Transgender Female | 1 | 1 | 2
  Additional sex or gender | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 23 | 45
  White | 4 | 6 | 10
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment
Description: We defined feasibility as the total number of patients approached in order to accrue the final study sample size of n=60.
Time Frame: Duration of recruitment phase (9 months)
Population: The analysis population for this outcome measure (feasibility of recruitment) is larger than the study population as we included all patients approached for screening (n=92) to reach our study sample (n=60).
Measure: Number; unit: participants
Groups:
- No Arm Assignment in Screening Phase: Participants approached for screening and eligibility are not linked to the participants who enrolled and were eventually randomized to 1 of the 2 study arms.
Arm/Group | No Arm Assignment in Screening Phase
Number analyzed (Participants) | 92
participants | 92

2. Primary Outcome: Client Acceptability
Description: Client acceptability will be assessed via the Client Satisfaction Questionnaire-8 (CSQ-8). The CSQ-8 is an 8-item questionnaire, with a minimum value of 8 and a maximum score of 32. A higher score indicates greater client acceptability.
Time Frame: At treatment exit (approximately 9 months post-baseline)
Population: Client acceptability was only measured for participants in the CETA arm since this outcome reflects their overall satisfaction with the intervention. This population includes the 25 participants who completed the exit interview ~9 months post-baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CETA Protocol: Adapted Common Elements Treatment Approach (CETA): The intervention is a transdiagnostic cognitive behavioral therapy approach to treating any combination of depression, anxiety, post-traumatic stress, or substance use disorder that has been adapted the needs of adults with HIV and to additionally address HIV care engagement.
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 25 | 0
units on a scale | 29.3 (3.0) |

3. Primary Outcome: Fidelity
Description: Counselor fidelity to CETA will be rated by the trainer based on the trainer's supervisory experience working with CETA counselors. After all CETA patients complete the study, the trainer will rate up to 5 cross-cutting aspects of CETA delivery and 13 CETA components targeting specific symptoms for fidelity. The trainer will rate the degree of confidence on a scale of 0 ("Not at all") to 4 ("Completely") that the counselor was routinely delivering each cross-cutting aspect or component of CETA with fidelity, for those aspects and components that the trainer had experience supervising the counselor in. The fidelity rating will be calculated separately for the 2 CETA counselors and reported as the mean score across the number of CETA aspects and components rated by the trainer. Higher scores indicate greater fidelity to CETA.
Time Frame: At the end of CETA completion or withdrawal, across all CETA participants
Population: The analysis population includes the total number of clients assigned to each counselor.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CETA Counselor 1: CETA counselor # 1
- CETA Counselor 2: CETA Counselor #2
Arm/Group | CETA Counselor 1 | CETA Counselor 2
Number analyzed (Participants) | 24 | 6
units on a scale | 3.3 (0.72) | 3.0 (0)

4. Secondary Outcome: Number of Participants Suppressed HIV RNA Viral Load
Description: HIV RNA viral load <200 copies/mL
Time Frame: 4 months post-baseline
Population: The analysis population includes all participants with a collected 4-month viral load.
Measure: Count of Participants; unit: Participants
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 21 | 27
Participants | 13 | 18

5. Secondary Outcome: Number of Participants With Suppressed HIV RNA Viral Load
Description: HIV RNA viral load <200 copies/mL
Time Frame: 9 months post-baseline
Population: This analysis population includes all participants with a completed viral load at 9 months post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 24 | 26
Participants | 17 | 17

6. Secondary Outcome: HIV Appointment Attendance
Description: Health Resources and Services Administration (HRSA) attendance measure: Engaged in care if attended >=2 HIV primary care visits >= 90 days apart in the 12 months after baseline.
Time Frame: From baseline to 12 months post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 30 | 30
Participants | 22 | 22

7. Secondary Outcome: Depressive Symptoms
Description: Patient Health Questionnaire-9 (PHQ-9) score; minimum score is 0, maximum score is 27, with higher scores meaning a worse outcome.
Time Frame: 4 months post-baseline
Population: The analysis population includes all participants with a completed interview at 4 months post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 27 | 28
score on a scale | 11.1 (6.8) | 9.8 (6.9)

8. Secondary Outcome: Anxiety Symptoms
Description: Generalized Anxiety Disorder-7 (GAD-7) anxiety subscale score; minimum score is 0, maximum score is 21, with higher scores meaning a worse outcome.
Time Frame: 4 months post-baseline
Population: The analysis population includes all participants with a completed interview at 4 months post-baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 27 | 28
score on a scale | 10.4 (5.4) | 9.3 (5.9)

9. Secondary Outcome: Post-traumatic Stress Symptoms
Description: PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5); minimum score is 0, maximum score is 80, with higher scores meaning a worse outcome.
Time Frame: 4 months post-baseline
Population: The analysis population includes all participants with a completed interview at 4 months post-baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 27 | 28
score on a scale | 33.7 (19.2) | 28.9 (17.3)

10. Secondary Outcome: Substance Use Symptoms
Description: The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST); each substance is scored separately. The minimum score is 0, maximum score is 39, with higher scores meaning a worse outcome. For this outcome, we will report substance use symptoms at 4 months post-baseline for the substance with the highest score at baseline only.
Time Frame: 4 months post-baseline
Population: The analysis population includes all participants with a completed interview at 4 months post-baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 27 | 28
score on a scale | 10.0 (8.1) | 7.9 (7.5)

11. Secondary Outcome: HIV Kept Visit Attendance
Description: Mean kept visit proportion: Total number of kept visits HIV clinical care visits divided by total number of missed plus kept HIV clinical care visits.
  For one individual: The numerator in this proportion is all the scheduled HIV clinical care visits a participant attended from baseline to 12-months post-baseline.The denominator in this proportion is all the scheduled HIV clinical care visits a participant attended plus all the scheduled HIV clinical care visits a participant did not attend or 'missed' from baseline to 12-months post-baseline.
  For each arm: We calculated the mean kept visit proportion per study arm by adding each individual kept visit proportion and dividing by the total number of participants in each arm.
Time Frame: From baseline to 12 months post-baseline
Population: Analysis population includes all participants with data on their total number of HIV care visits collected from baseline to 12 months post-baseline.
Measure: Mean (Standard Deviation); unit: Proportion of HIV care visits
Arm/Group | CETA Protocol | Enhanced Usual Care
Number analyzed (Participants) | 28 | 30
Proportion of HIV care visits | 0.74 (0.27) | 0.70 (0.27)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time a participant provided informed consent and was randomized in the study through ~ 12 months post-randomization.
Description: We collected systematic information on serious adverse events via a study collection form.
Arm/Group | CETA Protocol | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT04163341/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT04163341/ICF_001.pdf